CLINICAL TRIAL: NCT06871501
Title: "Observational, Retrospective and Prospective, Non-interventional, Multicentre National Registry-based Study to Collect Information on the Use of Genomic Testing in the Management of Early Stage HR+/HER2- Breast Cancer"
Brief Title: "Observational, Retrospective and Prospective, Non-interventional, Multicentre on the Use of Genomic Testing in the Management of Early Stage HR+/HER2- Breast Cancer"
Acronym: GIM29-GIMOMIC
Status: Not yet recruiting | Type: Observational
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Other Study IDs: GIM29-GIMOMIC
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Genomic testing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective cohort: For prospective cohort: genomic tests will be performed on all patients who meet the criteria for access to testing as set out in the Ministerial Decree of 18/05/2021, unless otherwise agreed by the reference Breast Unit, in accordance with the specific diagnostic pathways activated by each site.
- Retrospective cohort: For retrospective cohort: data for patient referred for genomic testing following Ministerial Decree 18/05/2021 will be collected. The retrospective cohort will contribute to expanding our knowledge of the clinico-pathological characteristics of patients who underwent genomic testing. This comprehensive understanding of the clinico-pathological profile of patients undergoing genomic testing will enable a more thorough assessment of the clinical dynamics and therapeutic decisions associated with genomic testing results, including the analysis of their possible evolution over the years.

SUMMARY:
The study aims to establish an Italian registry for the implementation of the use of genomic tests in patients with HR +/HER2- breast cancer at intermediate risk of recurrence after the entry into force of the Ministerial Decree of 18/05/2021. The decree has established the reimbursability of genomic testing for breast cancer patients, thereby influencing clinical decision-making and patient management within Breast Units. In addition, the study aims to evaluate the clinical impact of the use of genomic testing on the type of adjuvant treatment, in terms of change of treatment indication by breast units according to the test result.

DETAILED DESCRIPTION:
The study is a retrospective and prospective, non-interventional, observational registry-based study that will enroll all patients with ER +/HER2-negative, T1-3 breast cancer with negative axillary lymph nodes or up to 3 positive axillary lymph nodes for whom Breast Units require genomic test to support adjuvant therapy decisions, according to current clinical practice. For prospective cohort: genomic tests will be performed on all patients who meet the criteria for access to testing as set out in the Ministerial Decree of 18/05/2021, unless otherwise agreed by the reference Breast Unit, in accordance with the specific diagnostic pathways activated by each site. For retrospective cohort: data for patient referred for genomic testing following Ministerial Decree 18/05/2021 will be collected. The patient's baseline demographic characteristics, tumor clinicopathological features, pre and post-test therapeutic indication (CET vs ET), the test results, the actual adjuvant treatment received and time around data will be recorded in a dedicated registry.

ELIGIBILITY:
Inclusion Criteria:

1. . Age ≥ 18 years
2. PS ECOG 0-1
3. Histologically confirmed early breast carcinoma with positivity for hormone receptors (ER+ IHC >10%) and HER2 negative (IHC value 0 1+ and/or FISH not-amplified)
4. Primary resective surgery for early breast cancer with adequate assessment of lymph node status (sentinel lymph node biopsy or complete axillary dissection), with one of the following diagnostic stages:

   * T1-3, N0, M0
   * T1-3, pN1mic, M0
   * T1-3, pN1a, M0
5. Indication for adjuvant treatment with endocrine therapy (ET) or chemo endocrine therapy (CET), according to the decision of the reference Breast Unit
6. Meeting the criteria for "intermediate" risk, i.e., no "low" or "high" risk of recurrence, as defined in the ministerial decree of 18/05/21:

   * Low risk defined by at least 5 of the following: G1, T1a-b, KI67 < 15, N neg, ER > 80%
   * High risk, defined by at least 4 of the following: G3, T > 2, Ki67 > 30, N pos, ER < 30%
7. Indication for genomic test (Oncotype DX®, Mammaprint®, PAM50 Prosigna®, Breast Cancer Index®, EndoPredict®) by the Breast Unit
8. Ability to provide written informed consent to participate in the registry study, approved by the local Ethics Committee.
9. The patient underwent genomic testing starting from September 2021

Exclusion Criteria:

1. Low-risk and High-risk patients as defined in the Ministerial Decree of 18/05/21
2. ER negative and/or HER2 positive tumours
3. More than 3 lymph nodes involved at clinical/pathological staging
4. Invasive tumours <2mm evaluated by local pathologists
5. Previous history of breast cancer
6. Synchronous breast cancers
7. Multifocal tumours
8. Metastatic disease
9. Contraindications to adjuvant treatments
10. Performance status (PS ECOG) > 1 and / or other clinical factors that would make the patient a candidate and unsuitable for systemic adjuvant treatment or have received an exclusive indication for precautionary hormone therapy as part of the Breast Unit collegial assessment.
11. Psychiatric diagnosis that may affect the ability to participate in this study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study is a retrospective and prospective, non-interventional, observational registry-based study that will enroll all patients with ER +/HER2-negative, T1-3 breast cancer with negative axillary lymph nodes or up to 3 positive axillary lymph nodes for whom Breast Units require genomic test to support adjuvant therapy decisions, according to current clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Establishment of a prospective Italian observational registry for the implementation of genomic tests in patients with HR +/HER2- breast cancer | Until November 2026
  Establishment of a prospective Italian observational registry for the implementation of genomic tests in patients with HR +/HER2- breast cancer at intermediate risk of recurrence after the adoption of the Ministerial Decree of 18/05/2021
Measurement of the impact of genomic testing on adjuvant treatment choice (CET vs ET only) | Until November 2026
  Rate of adjuvant treatment choice's change following the genomic test result (Breast Unit's pre-test vs post-test indication)
Measurement of the impact of genomic testing on adjuvant treatment choice (CET vs ET only) | Until November 2026
  Saving in adjuvant chemotherapy compared to the pre-test indication
Measurement of the impact of genomic testing on adjuvant treatment choice (CET vs ET only) | Until November 2026
  Addition of adjuvant chemotherapy to endocrine therapy alone compared to the pre-test indication
Measurement of the impact of genomic testing on adjuvant treatment choice (CET vs ET only) | Until November 2026
  Type of adjuvant treatment the patient actually received

SECONDARY OUTCOMES:
Record the predominant demographic and clinical characteristics of the patients for whom genomic testing was indicated. | Until November 2026
  Record the predominant demographic and clinical characteristics of the patients for whom genomic testing was indicated.
Describe which genomic tests are used and the factors involved in the selection of genomic tests. | Until November 2026
  Describe which genomic tests are used and the factors involved in the selection of genomic tests.
Identify any inequalities in access to the genomic tests in different geographical areas of the country. | Until November 2026
  Identify any inequalities in access to the genomic tests in different geographical areas of the country.
Analyse the prescriptive adequacy and the compliance | Until November 2026
  With the inclusion criteria for genomic tests.
Record the distribution of demographic and clinical characteristics in the group of patients with changed treatment recommendation compared to the group of patients with unchanged indication after genomic test. | Until November 2026
  patient age comorbidities, tumour size, number of positive lymph nodes, tumour grade
Evaluate the impact of the test on the timing of activation of adjuvant treatment | Until November 2026
  Time from diagnosis to request for genomic test
Evaluate the impact of the test on the timing of activation of adjuvant treatment | Until November 2026
  Time from request for the genomic test to result
Evaluate the impact of the test on the timing of activation of adjuvant treatment | Until November 2026
  Time from test result to activation of adjuvant chemotherapy, if indicated
Evaluate the impact of the test on the timing of activation of adjuvant treatment | Until November 2026
  Time from diagnosis to activation of adjuvant chemotherapy, if indicated

CONTACTS AND LOCATIONS:
Locations (25):
- Italy (25):
  - A.O. San Giuseppe Moscati, Avellino, AV
  - Ospedale Papa Giovanni XXIII, Bergamo, BG
  - Policlinico S. Orsola-Malpighi, Bologna, BO
  - Spedali Civili di Brescia, Brescia, BS
  - Asrem - Azienda Sanitaria Regionale del Molise, Termoli, CB
  - Azienda Ospedaliera" Sant'Anna e San Sebastiano", Caserta, CE
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Azienda Ospedaliero-Universitaria Arcispedale S. Anna, Ferrara, FE
  - Azienda Ospedaliera Universitaria Careggi, Florence, FI
  - IRCCS Ospedale Policlinico San Martino, Genova, GE
  - IRCCS Ospedale San Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - IRCCS Humanitas Research Hospital, Rozzano, MI
  - IRCCS Centro di Riferimento Oncologico (C.R.O.), Aviano, PD
  - Ospedale S. Stefano, Prato, PO
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE
  - Istituto Nazionale Tumori Regina Elena, Roma, RM
  - Ospedale Infermi di Rimini, Rimini, RN
  - Ospedale San Bortolo di Vicenza, Vicenza, VI
  - A.O.R.N. "A. Cardarelli", Napoli
  - AORN - Ospedali dei Colli, Napoli
  - Azienda Ospedaliero Universitaria Federico II, Napoli
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - A.O.U. Maggiore della Carità di Novara, Novara
  - P.O."Santa Maria delle Grazie" di Pozzuoli, Pozzuoli

DOCUMENTS (1):
  • Study Protocol (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT06871501/Prot_000.pdf